CLINICAL TRIAL: NCT03225690
Title: Does Preemptive Epidural Morphine Prevent Remifentanil Induced Hyperalgesia
Brief Title: Prevention of Hyperalgesia With Epidural Morphine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Dr, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hyperalgesia
Record Dates: First submitted 2017-06-02; First posted 2017-07-21 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2017-11

CONDITIONS: Hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- serum physiologic (Placebo Comparator): 2 ml serum physiologic will apply via epidural catheter before surgical incision.
  Interventions: Drug: Serum physiologic
- Preemptive Morphine (Active Comparator): 1 mg morphine will apply via epidural catheter before surgical incision.
  Interventions: Drug: Morphine
- Morphine (Active Comparator): 1 mg morphine will apply via epidural catheter before at the time point of the peritoneum closed.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Prevention of remifentanil induced hyperalgesia
  Other Names: Group I-II
  Arms: Morphine; Preemptive Morphine
Drug: Serum physiologic — For placebo, serum physiologic will use
  Other Names: Group III
  Arms: serum physiologic

SUMMARY:
American Society of Anaesthesiologist physical status (ASA) I-III 105 patients who undergoing major abdominal surgery in obstetric and gynaecology clinic were recruited to this study. Patients were randomized into the 3 groups. Lumbar epidural catheter will be inserted to the all patients. After than anaesthesia induction will provide with 2 mg/kg propofol and 0.6 mg/kg rocuronium. Desflurane and azot protoxit (N2O)-O2 will use for anaesthesia maintenance. During surgical operation, 0.3 microgram/kg/h remifentanil infusion will continuous till the end of surgery. In group I, 2 ml serum physiologic (0.9 NaCL)will apply from epidural catheter before surgical incision. In group II, 1 mg morphine will apply from epidural catheter before surgical incision. In group III, 1 mg morphine will apply from epidural catheter at the time point of peritoneum is closed. Epidural patient controlled analgesia will provide with bupivacaine for postoperative analgesia. Postoperative pain will be assessed with numerical pain scale. Postoperative analgesic requirement will be calculated. Hyperalgesia will detect with algometer and von Frey ligaments.

DETAILED DESCRIPTION:
This randomized, double blind, controlled study will perform after obtaining informed consent and ethics approval. American Society of Anaesthesiologist physical status (ASA) I-III 105 patients who undergoing major abdominal surgery in obstetric and gynaecology clinic were recruited to this study. Patients were randomized into the 3 groups with computerized randomization programme. Lumbar epidural catheter will be inserted to the all patients. After than anaesthesia induction will provide with 2 mg/kg propofol and 0.6 mg/kg rocuronium. Desflurane and N2O-O2 will use for anaesthesia maintenance. During surgical operation, 0.3 microgram/kg/h remifentanil infusion will continuous till the end of surgery. In group I, 2 ml serum physiologic (0.9 NaCL)will apply from epidural catheter before surgical incision. In group II, 1 mg morphine will apply from epidural catheter before surgical incision. In group III, 1 mg morphine will apply from epidural catheter at the time point of peritoneum is closed. Epidural patient controlled analgesia will provide with bupivacaine for postoperative analgesia. Postoperative pain will be assessed with numerical pain scale. Postoperative analgesic requirement will be calculated. Hyperalgesia will detect with algometer and von Frey ligaments.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* Patients who undergoing major abdominal surgery

Exclusion Criteria:

* ASA IV and up
* Coagulopathy

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesic requirement | Till the postoperative 24th hour.
  Calculation of epidural bupivacain consumption

SECONDARY OUTCOMES:
Algometer values | Till the postoperative 24th hour.
  Postoperative pain will detect with algometer

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Biricik, Study Chair — Cukurova University
Locations (1):
- Çukurova University Balcalı Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No